CLINICAL TRIAL: NCT05342883
Title: Pilot Study of Resection and GammaTile Followed by Concomitant External Beam Radiation Therapy (EBRT) and Temozolomide (TMZ) and Adjuvant in Newly Diagnosed Glioblastoma (GBM)
Brief Title: GammaTile and Stupp in Newly Diagnosed GBM
Acronym: GESTALT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-103
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Newly Diagnosed; Stupp; GammaTile; External Beam Radiation Therapy; Temozolomide; Resection; Brain; Tumor; EBRT; Glioma
MeSH Terms: conditions — Glioblastoma; Neoplasms; Glioma

STUDY DESIGN:
Intervention Model Description: The intervention is the addition of GammaTile radiation therapy to the standard of care Stupp Protocol treatment of newly diagnosed GBM patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: Resection, GammaTile and Stupp Protocol (Other): Resection, Gamma Tile and Stupp Protocol
  Interventions: Device: Surgical tumor resection, GammaTile radiation therapy implantation, Stupp protocol (EBRT and Temozolamide)

INTERVENTIONS:
Device: Surgical tumor resection, GammaTile radiation therapy implantation, Stupp protocol (EBRT and Temozolamide) — At the initiation of the surgical phase maximal safe resection will be undertaken, and after 25 + 4 from surgery participants will start the concomitant phase and receive daily temozolomide (TMZ, 75mg/m2) and 20 fractions external beam radiation (EBRT). The EBRT treatment will be to the operative bed and any residual disease identified at the time of the imaging obtained for EBRT planning. The EBRT planning will utilize the GT implant dosimetry with the intent that the dose received from the GT will be accounted for during the EBRT treatment planning process. Twenty-eight days ±7 after the completion of concomitant TMZ and EBRT, participants will enter the adjuvant phase and will be treated with TMZ (150-200mg/m2) for 5 days at the start of every 28- day cycle, for 6 cycles.

SUMMARY:
In summary, standard of care postoperative chemoradiation for patients with newly diagnosed GBM does not routinely provide durable local control or prolonged overall survival. As discussed above it seems unlikely that patient outcomes will be significantly improved with radiation dose escalation given at the time of the EBRT boost. However, as most failures are local, improving LC could potentially improve the OS of patients. To do this, we propose a shift in the traditional radiation paradigm. This study will assess the feasibility and tolerability of adding GT radiation therapy as an upfront boost at the time of maximum safe resection, along with the backbone of the current standard of care approach, concomitant and adjuvant temozolomide +/- TTF, for patients with newly diagnosed GBM. GT, a novel brain brachytherapy device utilizing Cs-131 embedded in bioresorbable collagen tiles, offers a more sophisticated carrier and a shorter half-life radioisotope, Cs-131. Use of this device allows for radiation initiation at an earlier time point and a more rapid dose delivery and possibly more effective tumor control particularly for rapidly proliferating tumors such as GBM. Two prospective studies have demonstrated the safety and efficacy of re-irradiation with GT in patients with recurrent GBM. The overarching goal of this single-arm, open label phase 4 study is to determine the feasibility and tolerability of treating patients with GammaTile in combination with the Stupp Protocol and how to proceed with testing this treatment in a future, larger, randomized clinical study. The aims of the study are to demonstrate that the use of GammaTile at the time of surgery is well tolerated and does not delay the start of the Stupp protocol. Efficacy outcomes (e.g., LC, OS, PFS) will also be described.

DETAILED DESCRIPTION:
This study seeks to explore if GT, given its unique radiobiological and physical characteristics, may permit safe dose escalation and intensification and thereby provide a benefit to newly diagnosed GBM patients in terms of OS and LC when incorporated into the framework of the Stupp protocol. In this study, GT is utilized as an upfront boost at the time of maximum safe resection and dosimetrically integrated into what is otherwise standard of care therapy.

Patients in this study will receive doses from two different forms of radiation treatment, initially from Cs-131 BT with GT and subsequently from fractionated EBRT. In order to ensure both patient safety and adequacy of treatment, we have chosen to stipulate and evaluate the coverage of the tumor volumes and OARs using the doses combined from both these treatments. The intention is that with this methodology the doses received by the target volumes and relevant OARs from the implanted Cs-131 will be accounted for during EBRT treatment planning. This dose combination, accomplished using radiobiological modeling, is frequently undertaken in breast, prostate, and gynecological malignancies. To provide oversight and planning feedback, the first three patients enrolled at each site will undergo review by the Clinical Oversight Committee (COC) at two points for each patient, once after the GT implant, and before starting EBRT treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be ≥ 18 years of age
2. Histopathological and molecular confirmation of newly diagnosed GBM using IDH mutation testing (such as immunohistochemistry for IDH1 R132H) must be performed as part of SOC. A central lab will perform cytogenetics testing. Note: In patients without prior biopsy, diagnosis will be suspected preoperatively, but must be confirmed by molecular testing (i.e., must be IDH wild type). Patients with confirmed pathology from biopsy prior to enrollment are able to participate if they meet all other study requirements. Enrolled patients not ultimately confirmed to have molecular GBM or are found to have IDH mutated tumors after resection and GT placement (if appropriate), will be followed for safety. If tested before screening, patients known to have IDH mutated tumors should not be invited to participate or consented/enrolled.
3. Adequate tissue for central submission to determine methylation promoter status. Patients with either methylated or unmethylated MGMT promoter status are included, and this status must be confirmed by central pathology review. Note: Patients with tissue that is insufficient or inadequate for analysis, fails MGMT testing, or has indeterminate MGMT promoter status will receive GT (if indicated) and will be part of the ITT/safety population but will be excluded from the PP population analyses.
4. A supratentorial tumor that in the opinion of the enrolling neurosurgeon is a) amenable to attempted gross total resection (GTR) and b) has a maximum preoperative diameter of 6 cm or less when considering all tumor planned for resection (enhancing and non-enhancing). If multifocal, must be fully resectable in one operative bed. Prior diagnostic biopsy allowed. Surgical protocol will follow current institutional standards. If intraoperative MRI is utilized, details will be captured.
5. Able to receive 5-aminolevulinic acid (5-ALA, Gleolan) or other institutionally standard immunofluorescent-guidance such as fluorescein, prior to surgery to optimize GTR of enhancing tumor.
6. Patient is appropriate candidate to receive SOC treatment for newly diagnosed GBM as usually practiced (Stupp protocol with at least 6 cycles and up to 12 cycles of TMZ).
7. Concomitant systemic or local anti-cancer medications or treatments are prohibited in this study (with the exception of TTF) before progression.
8. Anti-angiogenic therapy (e.g., bevacizumab and its biosimilars) or steroid use is allowed for symptom management (e.g., brain edema or symptomatic pseudoprogression) as per institutional standard. Note: For both agents, utilization of the lowest useful doses and shortest useful courses are encouraged. At failure, tumor therapeutic dose of anti-angiogenic therapy (e.g., bevacizumab and its biosimilars) or other therapies can be utilized for treatment at the investigators' discretion.
9. Karnofsky Performance Scale (KPS) score of ≥ 70.
10. Eastern Cooperative Oncology Group Performance Score (ECOG-PS) of 0-2.
11. Ability to understand and the willingness to sign (personally or by a legally authorized representative) the written IRB approved informed consent document prior to performance of any study-related procedures.
12. Ability to understand English or Spanish.
13. Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests and accessible for follow-up after treatment termination.
14. Men and women of childbearing potential must be willing to employ adequate contraception throughout the study and for men for up to 3 months after completing treatment.
15. Satisfactory hematology as evidenced by standard pre-surgery labs:

    1. Hemoglobin ≥ 10 g/dl
    2. Leukocytes ≥ 2,000/mm3
    3. Absolute neutrophil count (ANC) ≥ 1,500/mm3
    4. Platelets ≥ 100,000/mm3
    5. Total bilirubin ≤ 2.0 x institutional/lab upper limit of normal (ULN)
    6. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) ≤ 2.5 x ULN
    7. Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN
    8. Serum creatinine ≤ 1.5 x ULN OR creatinine clearance (CrCl) ≥ 50mL/min (if using the Cockcroft-Gault formula)
    9. Absolute lymphocyte count between 1,000 and 4,800 per microliter of blood.

Exclusion Criteria:

1. Known to be IDH mutated glioma by prior biopsy.
2. Patients not appropriate for concomitant or maintenance temozolomide.
3. Previous chemotherapy or radiotherapy to the head or neck region resulting in overlapping fields or prior surgery to the brain to resect other brain tumors.
4. Staged surgery planned (prior biopsy allowed).
5. Bilateral tumors, or multi-focal tumors that cannot be encompassed in one operative field.
6. Enhancing extension into brainstem or thalamus, or significant invasion into the corpus callosum that would preclude a high likelihood of GTR.
7. Prior invasive malignancy (except non-melanomatous skin cancer, cervical cancer in situ) unless disease free for a minimum of 2 years
8. Definitive clinical or radiologic evidence of cancer outside the brain (excluding nonmelanomatous skin cancer, or other types of indolent cancers) not needing active treatment within the past 2 years. Contact the Medical Monitor to review any inquiries on indolent cancers allowed.
9. Concomitant systemic or local anti-cancer medications or treatments in use or planned (with the exception of TTF before progression or on protocol TMZ).
10. Planned use of adjuvant anti-angiogenic therapy (e.g., bevacizumab and its biosimilars) specifically for tumor treatment
11. Enrollment in another investigational study or planned use of investigational therapies. Note: Experimental therapies or enrollment in a subsequent study are allowed after a patient on study has a local recurrence or distant brain failure.
12. Patients with contraindication to MRI or CT
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide, bovine -derived collagen, 5-ALA or other institutionally standard immunofluorescent-guidance compounds, such as fluorescein.
14. Participants with severe intercurrent illness that will prohibit subsequent chemotherapy and radiotherapy including, but not limited to, unstable systemic disease including ongoing or active infection, COVID-19, uncontrolled hypertension, serous cardiac arrythmia requiring medication, acute cardiovascular disease or clinically manifested myocardial insufficiency or history of myocardial infarction during the past 6 months prior to screening, severe psychiatric illness or other illness that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with proper assessment of safety and adverse events of the prescribed regimens.
15. Women who are pregnant or lactating. Women of child-bearing potential must have a negative urine test or serum beta human chorionic gonadotrophin (b-HCG) documented no greater than 14 days prior to study registration unless they are surgically sterile (e.g. oophorectomy, hysterectomy, tubal ligation) or menopausal. Menopause is defined as 12 months of amenorrhea in a woman over 45 in the absence of possible causes for amenorrhea (e.g., low body fat, hormonal imbalances, etc.)
16. Any concomitant therapy (e.g., strict ketogenic diet, high dose vitamin C) that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of any of the study treatments.
17. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent.
18. Participants who, in the investigator's opinion, are unable to understand the protocol or to give informed consent (personally or by a legally authorized representative), have a history of poor cooperation, noncompliance with medical treatment, or difficulty in returning for follow up care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in the Intent to Treat (ITT) population who were able to start the Concomitant Phase (start is defined as first day of EBRT) between 21 and 35 days postoperatively. | 21-35 days
  Feasibility of using GammaTiles in patients who will also be treated with the Stupp Protocol.
Overall incidence of treatment related (possibly, probably, or definitely) grade ≥3 (CTCAE v5) adverse events in the safety analysis (ITT) population. | 24 months
  Safety of treating patients treated with GammaTiles in addition to the Stupp protocol.

SECONDARY OUTCOMES:
Percentage of patients in the per protocol (PP) population who were able to start the Concomitant Phase (start is defined as first day of EBRT) between 21 and 35 days postoperatively. | 21-35 days
  Feasibility of using GammaTiles in patients who will also be treated with the Stupp Protocol.
Incidence of treatment related (possibly, probably, or definitely) grade ≥3 (CTCAE v5) adverse events during each phase (surgical phase, concomitant phase, and adjuvant phase, in both the safety analysis (ITT) and PP populations. | 24 months
  Secondary safety endpoint-assessment of safety in those patients who were treated per protocol
Percentage of pre-screened patients consenting to participate in the study. | Pre-Screening to Consent
  Assessment of ease of enrollment.
Percentage of patients lost to attrition after consenting to participate. | up to 24 months
  Assessment of attrition

OTHER OUTCOMES:
Safety (Complications and Adverse Events) | 24 months
  Complications can occur with any neurosurgical procedure and include but are not limited to problems with wound healing, cerebrospinal fluid leaks, infection, acute or delayed hemorrhage, seizures, and adhesion formation. EBRT complications can include but are not limited to nausea, vomiting, alopecia, skin toxicity, vertigo, problems with attention or concentration, worsening neurological symptoms, and radionecrosis of brain and non-brain tissues.
Overall Survival | 12,18 and 24 months
  For this feasibility study, median overall survival, and overall survival at 12, 18 and 24 months will be analyzed in both the ITT and per protocol population.
Progression Free Survival | 24 months
  Progression Free Survival (PFS) is defined as time from the date of surgery to date of progression, death, or last known follow-up (censored).
Karnofsky Performance Status Scale | 24 months
  The Karnofsky Performance Status Scale is used to assess functional impairment. Score 0 to 100, with 100 being no impairment of performance
Eastern Cooperative Oncology Group Performance Status Scale | 24 months
  The Eastern Cooperative Oncology Group Performance Status scale is a simple, 5 point scale that can be used in daily practice measure tp measure functional status. Scores of 0-5 with 0 being fully active, and 10 being dead.
Immune Competence | 24 months
  The immune system plays a major role in suppressing the development and growth of primary brain tumors. Therefore immune competence will also be measured by assessing absolute lymphocyte counts.
Toxicity Analysis Using Radiobiologically based BT Plus EBRT Dose Combinations | 24 months
  Systematic evaluation of the toxicity outcomes using this methodology is an exploratory objective of the study.
Immune competence, as measured by absolute lymphocyte counts (ITT and PP populations) | 24 months
  Assessment of the impact of therapy on immune competence.
Examine intracranial radiation toxicity outcomes in a population of patients for whom radiobiological modeling was used to combine dose of Cs 131 brachytherapy and EBRT (ITT and PP populations) | 24 months
  Assessment of the incidence of radiation toxicity

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - HonorHeath Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Keck Medicine of USC, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Advent Health Orlando, Orlando, Florida
  - Florida Health Sciences Center, Inc. d/b/a Tampa General Hospital, Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - RUSH University, Chicago, Illinois
  - Indiana University Office of Clinical Research, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis University Hospital Center, St Louis, Missouri
  - ECU Health Medical Center - Vidant, Greenville, North Carolina
  - Kettering Medical Center, Kettering, Ohio
  - Brown University Health, Providence, Rhode Island
  - UTHealth Houston | Memorial Hermann Health System, Houston, Texas

IPD SHARING:
Plan to Share IPD: No